CLINICAL TRIAL: NCT00031850
Title: A Randomized Trial Of Raloxifene Plus Zoladex For Prevention Of Breast Cancer
Brief Title: Raloxifene and Goserelin in Preventing Breast Cancer in Women With a Family History of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: NCRI-IBIS-RAZOR; CDR0000069233 (Registry Identifier: PDQ (Physician Data Query)); EU-20053; UKCCCR-IBIS-RAZOR; ISRCTN17775670
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Raloxifene Hydrochloride

INTERVENTIONS:
Drug: goserelin acetate
Drug: raloxifene

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of raloxifene and goserelin may be effective in preventing breast cancer.

PURPOSE: Randomized pilot study to study the effectiveness of combining raloxifene and goserelin in preventing breast cancer in women who have a family history of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the feasibility of raloxifene and goserelin versus no medical intervention in women at high genetic risk for developing breast cancer.
* Compare the incidence of adverse effects in patients treated with these regimens.
* Compare the effect of these regimens on bone density, biochemical markers of bone turnover, and lipid profiles in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive goserelin subcutaneously once every month and oral raloxifene daily for 6-12 months.
* Arm II: Patients are screened for breast cancer every 6 months. In both arms, patients undergo annual mammograms.

Quality of life is assessed at baseline and at 1, 3, 6, and 12 months.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 150 patients (75 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* High genetic risk of developing breast cancer defined as one or more of the following:

  * BRCA1 or BRCA2 germ-line mutation
  * First-degree relative of known BRCA1 or BRCA2 mutation carrier
  * Family with 4 or more relatives diagnosed with female or male breast cancer or ovarian cancer before the age of 60
  * Two first-degree relatives diagnosed with breast cancer before the age of 40
  * p53 germ-line mutation (classical Li-Fraumeni syndrome (LFS) only)
  * First-degree relative of a carrier in a family with classical LFS
  * Risk equivalent to any of the above confirmed by clinical geneticist
* No evidence of breast cancer by mammography

  * Suspicious lesions must be confirmed as non-malignant
* No prior breast cancer
* No prior prophylactic mastectomy
* No plan for alternative prevention measures within the next 12 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 30 to 45

Sex:

* Female

Menopausal status:

* Premenopausal (follicle-stimulating hormone in premenopausal range if not menstruating)

Performance status:

* Not specified

Life expectancy:

* More than 10 years (excluding breast cancer risk)

Hematopoietic:

* Not specified

Hepatic:

* Adequate liver function

Renal:

* Adequate renal function

Cardiovascular:

* No prior deep vein thrombosis

Pulmonary:

* No prior pulmonary embolism

Other:

* Not pregnant
* Fertile patients must use effective nonhormonal contraception
* No psychological disorder that would preclude study compliance
* No prior malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or cervical cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent hormonal therapy (e.g., oral contraception or hormone replacement therapy)

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* At least 30 days or 5 half-lives since prior investigational drugs
* No concurrent anticoagulants

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2000-03; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Howell, MD, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital NHS Trust, Manchester, England, United Kingdom